CLINICAL TRIAL: NCT00205400
Title: Comparison of Patient Outcomes Using Different Delivery Models of Anticoagulation Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M-1999-0280
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Anticoagulation; Thromboembolism
MeSH Terms: conditions — Thromboembolism

INTERVENTIONS:
Procedure: medical care delivery model

SUMMARY:
Hypothesis: Does the time spent within the target INR range differ when patients are managed by AMD or IT models of anticoagulation care?

Experimental Design: The 36-month trial enrolled 192 eligible patients currently receiving chronic warfarin therapy at the William S. Middleton Memorial VA Hospital. Consenting patients are enrolled and randomized to 1 of 2 groups: usual clinic care with face-to-face visits every 4 weeks (AMS model) or clinic visits every 3 months with interim laboratory visits and telephone follow-up every 4 weeks (IT model). At study conclusion, the amount of time the INR is within target range will be compared between the two groups. Thromboembolic and bleeding event rates, patient knowledge, quality of life and healthcare utilization will also be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* completion of >3 months of warfarin
* indefinite warfarin therapy

Exclusion Criteria:

* patients who currently receive >25% of INR determinations per year from local labs
* extended absences from VA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192
Dates: Start 1999-08; Primary Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Percent time in therapeutic range (TTR) using modified version of Rosendaal method

SECONDARY OUTCOMES:
Event rates for thromboembolism, hemorrhages, hospitalizations, urgent care visits, emergency department visits, triage calls, INRs greater than 6.0 and quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Christine Sorkness, Pharm D, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States